## Investigator Initiated Trial Proposal - Acrysof<sup>TM</sup> IQ Vivity<sup>TM</sup> Toric

Date: 24/12/21

*Title:* Visual outcomes following implantation of the Acrysof <sup>TM</sup> IQ Vivity<sup>TM</sup> Toric Extended Vision Intraocular Lens

Setting: LEC Eye Centre, Ipoh, Malaysia

**Background:** The Acrysof<sup>TM</sup> IQ Vivity<sup>TM</sup> is a new non-diffractive, UV-absorbing and blue light filtering hydrophobic aspheric intraocular lens (IOL) which has been reported to provide an extended range of vision from distance to near with a low incidence of visual disturbances. The toric version also compensates for corneal astigmatism.

*Objective:* The primary objective of this study is to evaluate the clinical outcomes following implantation of the Acrysof<sup>TM</sup> IQ Vivity<sup>TM</sup> Toric Extended Vision IOL. Secondary objectives will include level of spectacle independence as well as the tolerance to residual astigmatism or refractive error.

**Design:** This is a single-centre prospective interventional study of patients with significant cataract and subsequent bilateral implantations of the Acrysof<sup>TM</sup> IQ Vivity<sup>TM</sup> Toric Extended Vision IOL. All eyes will have a refractive target of emmetropia with the IOL power which provides the first myopic target closest to emmetropia selected for implantation. Visual outcomes will be assessed up to 3 months after surgery. Target sample size will be 60 eyes of 30 patients.

Primary outcome measures at 3 months:

- 1. Binocular uncorrected distance, intermediate (66cm) and near (40cm) acuities. Visual acuity scores will be converted to logMAR for analysis.
- 2. VF-14 Quality of Life questionnaire
- 3. Questionnaire for Visual Disturbance (QUVID)

#### Secondary outcome measures:

- 1. Uncorrected distance, intermediate (66cm) and near (40cm) acuities
- 2. Best corrected distance acuity, distance corrected intermediate acuity and distance corrected near acuity
- 3. Monocular and Binocular Defocus Curve
- 4. Refractive predictability and stability
- 5. Rotational stability of IOL
- 6. Vector analysis of astigmatic correction
- 7. Mesopic and photopic Contrast Sensitivity with CSV 1000

### **Inclusion Criteria:**

- Patients with visually significant cataracts in both eyes and significant pre-existing corneal astigmatism (as determined by the Barrett Toric Calculator) planned for phacoemulsification and implantation of Acrysof™ IQ Vivity™ Toric Extended Vision IOL
- Patients aged 18 years or older

#### **Exclusion Criteria:**

- Eyes with other ocular pathology which may significantly impact visual acuity (e.g. moderate to advanced age related macular degeneration, centre-involving diabetic maculopathy, moderate to advanced glaucoma, keratoconus, corneal dystrophy, etc)
- Eyes with amblyopia or strabismus
- Eyes with pre-existing zonular weakness or capsular compromise
- Eyes with intraoperative capsular rupture

- Eyes which had previously undergone refractive surgery

*Study Plan:* Study procedures will be conducted prospectively and results entered into a database created for the purpose of this study.

## Schedule of Visits:

| Procedure | Preop | Day 0 | POD 1 | POD 7 | POD 1m | POD 3m |
|----------------------------|-------|-------|-------|-------|--------|--------|
| Demographics | 1 | | | | | |
| Medical/Ocular History | 1 | | | | | |
| Manifest Refraction | √ | | | √ | √ | 1/ |
| UCVA | 1 | | 1 | 1/ | √ | 1/ |
| BCVA | 1/ | | | 1/ | 1/ | 1/ |
| Slit lamp examination | 1 | | √ | 1 | 1/ | 1/ |
| Dilated fundus examination | 1 | | | | 1/ | 1/ |
| Biometry | 1 | | | | | |
| IOL position | | | | 1 | 1/ | |
| VF-14 | | | | | | 1/ |
| Contrast Sensitivity | | | | | | 1/ |
| QUVID | | | | | 1/ | 1/ |
| Adverse Events | | 1/ | 1/ | 1 | 1/ | 1/ |

**Data Analysis:** Descriptive statistics will be computed using Microsoft Excel and astigmatic analysis will be done using the ASSORT calculator.

# Timeline and publication plan:

| Items | Estimated timelines |
|---|---|
| IRB Submission | July 2021 |
| Contracting | October 2021 |
| First Patient First Visit | October 2021 |
| Last Patient Last Visit | March 2022 |
| Data Processing and Analysis | April 2022 |
| Final Report | May 2022 |
| Publication plans | 3 <sup>rd</sup> quarter 2022 |
| Presentation plans | APACRS 2022, ESCRS 2022, AAO 2022, ASCRS |
| | 2023, APAO 2023 |